CLINICAL TRIAL: NCT06444178
Title: A Parallel Group Study in Healthy Participants to Quantitate Increases in Subclinical Gastrointestinal Blood Loss Following Administration of Aspirin Alone or in Combination With Rivaroxaban or Factor XI Inhibitors (REGN9933 or REGN7508)
Brief Title: Assessment of Gastrointestinal Blood Loss After Receiving Aspirin or Aspirin Plus Rivaroxaban, or Aspirin Plus REGN9933, or Aspirin Plus REGN7508 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R9933-HV-2424
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
Keywords: Gastrointestinal (GI) bleeding; Fecal occult blood testing (FOBT)
MeSH Terms: conditions — Hemorrhage | interventions — Aspirin; Rivaroxaban

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm 1: Aspirin (Active Comparator): Randomized 1:1:1:1
  Interventions: Drug: Aspirin
- Arm 2: Aspirin + REGN9933 (Experimental): Randomized 1:1:1:1
  Interventions: Drug: Aspirin; Drug: REGN9933
- Arm 3: Aspirin + REGN7508 (Experimental): Randomized 1:1:1:1
  Interventions: Drug: Aspirin; Drug: REGN7508
- Arm 4: Aspirin + Rivaroxaban (Active Comparator): Randomized 1:1:1:1
  Interventions: Drug: Aspirin; Drug: Rivaroxaban

INTERVENTIONS:
Drug: Aspirin — Oral administration
Drug: REGN9933 — Administered intravenous (IV)
  Arms: Arm 2: Aspirin + REGN9933
Drug: REGN7508 — Administered IV
  Arms: Arm 3: Aspirin + REGN7508
Drug: Rivaroxaban — Oral administration
  Arms: Arm 4: Aspirin + Rivaroxaban

SUMMARY:
This study is researching experimental drugs called REGN9933 and REGN7508 (called "study drugs") and comparing their effects to approved treatments of rivaroxaban and aspirin (called "standard treatments"). Aspirin will be given alone or in combination with the study drugs or the other standard treatments to look at their effects on blood loss in the intestines.

The aim of the study is to see if aspirin alone or the study drugs REGN9933 and REGN7508, when taken with aspirin, cause less minor intestinal bleeding than standard treatments rivaroxaban with aspirin.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index between 18.0 and 32.5 kg/m2 (inclusive) at the screening visit
2. Judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and electrocardiograms (ECGs) performed at screening and/or prior to administration of initial dose of study treatment
3. Normal aPTT, normal PT, and normal platelet counts at screening period and at the day 1 visit as defined by the local laboratory
4. Hemoglobin values within the normal range, per local laboratory, at the screening and day 1 visits
5. Negative FOBT at Baseline (visit 2) and visit 3 as defined in the protocol

Key Exclusion Criteria:

1. History of any major surgical procedure or clinically significant physical trauma in the last 6 months, in the opinion of the investigator, that may pose a risk to the participant by study participation
2. Whole blood donation within the previous 56 days or plasma donation within the previous 7 days prior to the screening visit
3. Hospitalized for any reason within 30 days of the screening visit
4. Estimated glomerular filtrate rate (eGFR) of <60 mL/min/1.73m2 at screening as described in the protocol.
5. Current smoker or former smoker, including e-cigarettes, who stopped smoking within 12 months prior to the screening visit
6. History of illicit drug or alcohol abuse within the last 2 years prior to the day 1 visit
7. Use of any prescription and nonprescription medications or nutritional supplements from approximately 2 weeks or 5 half-lives, as described in protocol
8. Has elective surgery planned to occur prior to end of study (EOS)

Note: Other Protocol Defined Inclusion/ Exclusion Criteria Apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Change in fecal hemoglobin content (FHC) | Baseline and up to day 22

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAE) | Up to day 100
Severity of TEAE | Up to day 100
Incidence of major bleeding | Up to day 100
Incidence of clinically relevant non-major (CRNM) bleeding | Up to day 100
Concentrations of REGN9933 | Up to day 29
Concentrations of REGN7508 | Up to day 29
Change in activated partial thromboplastin time (aPTT) | Baseline and up day 29
Change in prothrombin time (PT) | Baseline and up day 29
Incidence of Anti-drug antibody (ADA) to REGN9933 | Up to day 29
Titer of ADA to REGN9933 | Up to day 29
Incidence of ADA to REGN7508 | Up to day 29
Titer of ADA to REGN7508 | Up to day 29

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Fortrea Clinical Development, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/